CLINICAL TRIAL: NCT01445548
Title: Pilot Study of the Evaluation of Intravitreal Sirolimus in the Treatment of Bilateral Geographic Atrophy Associated With Age-Related Macular Degeneration
Brief Title: Sirolimus for Advanced Age-Related Macular Degeneration
Acronym: SIRGA2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110249; 11-EI-0249 (Registry Identifier: National Institutes of Health Clinical Center)
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2014-05

CONDITIONS: Age-Related Macular Degeneration; Geographic Atrophy
Keywords: Age-Related Macular Degeneration (AMD); Geographic Atrophy; Bilateral Geographic Atrophy; Sirolimus; Age Related Macular Degeneration; AMD
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus (Experimental): Participants initially received a 20 μL (440 μg) intravitreal injection sirolimus in the study eye at baseline and every two months thereafter unless contraindicated.
  As of September 2012, sirolimus intravitreal injections were no longer administered to participants.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus
  Other Names: Rapamune®; rapamycin

SUMMARY:
This study will determine whether a drug called sirolimus is safe to give to people with geographic atrophy (GA) and if it can help preserve vision in patients. GA is an advanced form of dry age-related macular degeneration (AMD). AMD affects the macula, the central part of the retina at the back of the eye needed for sharp, clear vision. There are two types of AMD, wet and dry. In dry AMD, cells in the macula die.

GA may be partially caused by inflammation. Sirolimus helps prevent inflammation and therefore may help people with GA. Researchers want to see whether sirolimus can help prevent vision loss in people with GA.

People at least 56 years of age who have GA related to AMD in both eyes may be eligible for this study.

This study requires at least 8 visits to the National Eye Institute over 1 year. Study visits will be every 2 months for 1 year.

Participants will undergo the following procedures:

* Participants will be screened with a medical history and physical exam. They will also have blood and urine tests, and eye exams. One eye will be selected as the study eye to receive the sirolimus injections.
* Participants will have a sirolimus injection into the study eye at the first visit and every 2 months thereafter unless contraindicated. There will be a follow-up eye exam 1 month after the first injection.

DETAILED DESCRIPTION:
Objective: Age-related macular degeneration (AMD), the leading cause of blindness in people over age 65 in the United States, is a heterogeneous clinical entity in which retinal degeneration occurs predominantly in the macula in the context of aging and leads to impairment of central visual acuity. AMD occurs in two general forms, one of which involves choroidal neovascularization (CNV) with subsequent formation of a disciform scar. This is often referred to as the neovascular or wet form. A second form, the subject of this study, is termed dry or atrophic macular degeneration and involves a constellation of clinical features that can include drusen, pigment clumping and/or retinal pigment epithelium (RPE) dropout and geographic atrophy (GA). GA can begin as a thinning of the RPE with involvement of the underlying choriocapillaris and subsequently lead to an atrophic change in the macula. Inflammation may play a role in the pathogenesis of GA. Sirolimus inhibits the production, signaling and activity of many inflammatory factors relevant to the development of GA. Therefore, the objective of this study is to investigate the safety and possible efficacy of serial sirolimus intravitreal injections in participants with bilateral GA.

Study Population: Six participants with bilateral GA associated with AMD will be enrolled. Initially, 10 participants with bilateral GA associated with AMD were to be enrolled. However, only six will be enrolled, as sirolimus intravitreal injections will no longer be administered to participants.

Design: In this single-center, prospective, controlled, unmasked, Phase I/II study, one eye of eligible participants was initially randomized to investigational product (intravitreal sirolimus) while the fellow eye was observed. Participants initially received a 20 μL (440 μg) intravitreal injection sirolimus in the study eye at baseline and every two months thereafter unless contraindicated. As of September 2012, sirolimus intravitreal injections were no longer administered to participants. Both the study and fellow eyes will be observed every two months until the study terminates. The study will not terminate until all participants have been followed through Month 12.

Outcome Measures: The primary outcome is the rate of change in area of GA based on masked grading by an external Reading Center of fundus photographs in the study eye and fellow eye at Month 12 compared to baseline. Secondary outcomes will include changes in best-corrected visual acuity (BCVA), changes in drusen area based on masked digital grading of fundus photography, absolute and relative changes in area of GA measured using fundus photography and autofluorescence imaging, and development of exudative AMD measured using optical coherence tomography (OCT). Safety outcomes will include the number and severity of adverse events (AEs). Ocular safety outcomes will be indicated by changes in visual acuity, ocular surface changes, intraocular inflammation and any other ocular changes not consistent with the natural progression of GA.

ELIGIBILITY:
Inclusion Criteria

1. 56 or older
2. Must understand and sign the protocol's informed consent document
3. Must have at least ½ disc area (approximately 1 mm^2) of GA compatible with AMD present in each eye

   GA is defined as one or more well-defined and often circular patches of partial or complete depigmentation of the RPE, typically with exposure of underlying choroidal blood vessels. Even if much of the RPE appears to be preserved and large choroidal vessels are not visible, a round patch of RPE partial depigmentation may be classified as early GA. The GA in each eye must be able to be photographed in their entirety, and it must not be contiguous with any areas of peripapillary atrophy, which can complicate area measurements
4. Must have at least one large druse (greater than or equal to 125 μm) in each eye
5. Must not have any evidence or history of exudative disease related to AMD in either eye as determined by a recent fluorescein angiogram performed within 4 months of study enrollment
6. Must have a steady fixation in both eyes in the foveal or parafoveal area and media clear enough for good quality photographs
7. Must have visual acuity of 20/400 or better in each eye
8. Female participants of childbearing potential and male participants able to father children must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent from intercourse, or agree to practice two acceptable methods of contraception throughout the course of the study and four months after their last study injection. Acceptable methods of contraception include:

   * hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring),
   * intrauterine device,
   * barrier methods (diaphragm, condom) with spermicide, or
   * surgical sterilization (hysterectomy or tubal ligation).

Exclusion Criteria

1. Actively receiving study therapy in another investigational study
2. Unable to comply with study procedures or follow-up visits
3. Evidence of an ocular disease other than AMD in either eye that may confound the outcome of the study (e.g., diabetic retinopathy with 10 or more hemorrhages or microaneurysms, uveitis, pseudovitelliform macular degeneration moderate/severe myopia)
4. Has any of the following: a) a history of macular laser, b) a history of photodynamic therapy (PDT), c) received an intravitreal injection of anti-vascular endothelial growth factor (VEGF) agent for wet/exudative AMD at any point, or d) received an intravitreal injection of any other agent (not an anti-VEGF agent) within four months prior to study enrollment

   Participants currently taking or who have previously taken AREDS vitamin supplementation are not excluded.
5. Has had a vitrectomy
6. Expected to need ocular surgery during the course of the trial
7. Has undergone lens removal in the last three months or yttrium aluminum- garnet (YAG) laser capsulotomy within the last month
8. On chemotherapy
9. On immunosuppressive medication
10. On ocular or systemic medications known to be toxic to the lens, retina or optic nerve
11. History of ocular herpes simplex virus (HSV)
12. Has a condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control)
13. Has a history of cancer (other than a non-melanoma skin cancer) diagnosed within the past five years
14. Has laboratory values outside normal limits and considered clinically significant by the investigator
15. Is currently taking one of the following drugs: amprenavir, atazanavir, clarithromycin, darunavir, delavirdine, erythromycin, fluconazole (at doses of 200mg or greater), fluvoxamine, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, posaconazole, quinupristin, ritonavir, saquinavir, telithromycin, troleandomycin, verapamil or voriconazole
16. Female participant is pregnant or breast-feeding.

Min Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wai T Wong, MD, PhD, Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Klein R, Klein BE, Jensen SC, Meuer SM. The five-year incidence and progression of age-related maculopathy: the Beaver Dam Eye Study. Ophthalmology. 1997 Jan;104(1):7-21. doi: 10.1016/s0161-6420(97)30368-6. PMID 9022098
- [Background] Klein R, Klein BE, Linton KL. Prevalence of age-related maculopathy. The Beaver Dam Eye Study. Ophthalmology. 1992 Jun;99(6):933-43. doi: 10.1016/s0161-6420(92)31871-8. PMID 1630784
- [Background] Edwards AO, Ritter R 3rd, Abel KJ, Manning A, Panhuysen C, Farrer LA. Complement factor H polymorphism and age-related macular degeneration. Science. 2005 Apr 15;308(5720):421-4. doi: 10.1126/science.1110189. Epub 2005 Mar 10. PMID 15761121
- [Result] Petrou PA, Cunningham D, Shimel K, Harrington M, Hammel K, Cukras CA, Ferris FL, Chew EY, Wong WT. Intravitreal sirolimus for the treatment of geographic atrophy: results of a phase I/II clinical trial. Invest Ophthalmol Vis Sci. 2014 Dec 18;56(1):330-8. doi: 10.1167/iovs.14-15877. PMID 25525171
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-EI-0249.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sirolimus
Started | 6
Completed | 5
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sirolimus
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.33 (8.45)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Rate of Change in Area of Geographic Atrophy (GA), Based on Masked, Digital Grading of Fundus Photography by an External Reading Center, in the Study Eye at 12 Months Compared to Baseline.
Time Frame: Baseline and Month 12
Population: The analysis was intention-to-treat (ITT). Although 6 participants were enrolled, only 5 were followed for 12 months.
Measure: Mean (Standard Deviation); unit: mm^2/month
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
mm^2/month | 0.19 (0.08)

2. Primary Outcome: Rate of Change in Area of Geographic Atrophy (GA), Based on Masked, Digital Grading of Fundus Photography by an External Reading Center, in the Fellow Eye at 12 Months Compared to Baseline.
Time Frame: Baseline and Month 12
Population: The analysis was intention-to-treat (ITT). Although 6 participants were enrolled, only 5 were followed for 12 months.
Measure: Mean (Standard Deviation); unit: mm^2/month
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
mm^2/month | 0.13 (0.06)

3. Secondary Outcome: Changes in Early Treatment Diabetic Retinopathy Study (ETDRS) Best-corrected Visual Acuity (BCVA) in the Study Eye at 12 Months Compared to Baseline
Description: Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20. One eye (the study eye) was initially randomized to receive intravitreal sirolimus and the fellow eye was observed as the control.
Time Frame: Baseline and Month 12
Population: The analysis was intention-to-treat (ITT). Although 6 participants were enrolled, only 5 were followed for 12 months.
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
ETDRS letters | -15.6 (7.23)

4. Secondary Outcome: Changes in Early Treatment Diabetic Retinopathy Study (ETDRS) Best-corrected Visual Acuity (BCVA) in the Fellow Eye at 12 Months Compared to Baseline
Description: as for outcome 3
Time Frame: Baseline and Month 12
Population: The analysis was intention-to-treat (ITT). Although 6 participants were enrolled, only 5 were followed for 12 months.
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
ETDRS letters | 0 (13.47)

5. Secondary Outcome: Absolute Change in Total Area of Macular GA, Based on Masked, Digital Grading of Fundus Photography by an External Reading Center, in the Study Eye at 12 Months Compared to Baseline.
Description: Geographic atrophy (GA) is the death of photoreceptors and surrounding cells in the retina. The death of these photoreceptors results in lesions that cause vision loss. The area of GA was determined using planimetry for color stereoscopic fundus images by masked graders at the Doheny Image Reading Center (University of Southern California, Los Angeles, CA).
  This outcome measure was calculated by subtracting the GA value for the study eye at baseline from the GA value for the study eye at Month 12.
Time Frame: Baseline and Month 12
Population: The analysis was intention-to-treat (ITT). Although 6 participants were enrolled, only 5 were followed for 12 months.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
mm^2 | 2.26 (0.94)

6. Secondary Outcome: Absolute Change in Total Area of Macular GA, Based on Masked, Digital Grading of Fundus Photography by an External Reading Center, in the Fellow Eye at 12 Months Compared to Baseline.
Description: as for outcome 5
Time Frame: Baseline and Month 12
Population: The analysis was intention-to-treat (ITT). Although 6 participants were enrolled, only 5 were followed for 12 months.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
mm^2 | 1.53 (0.75)

7. Secondary Outcome: Relative Change in Total Area of Macular GA, Based on Masked, Digital Grading of Fundus Photography by an External Reading Center, in the Study Eye at 12 Months Compared to Baseline.
Description: Geographic atrophy (GA) is the death of photoreceptors and surrounding cells in the retina. The death of these photoreceptors results in lesions that cause vision loss. The area of GA was determined using planimetry for color stereoscopic fundus images by masked graders at the Doheny Image Reading Center (University of Southern California, Los Angeles, CA).
  This outcome measure was calculated by dividing the absolute change in the total area of GA in the study eye at 12 months by the baseline value.
Time Frame: Baseline and Month 12
Population: The analysis was intention-to-treat (ITT). Although 6 participants were enrolled, only 5 were followed for 12 months.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
Ratio | 0.18 (0.09)

8. Secondary Outcome: Relative Change in Total Area of Macular GA, Based on Masked, Digital Grading of Fundus Photography by an External Reading Center, in the Fellow Eye at 12 Months Compared to Baseline.
Description: as for outcome 7
Time Frame: Baseline and Month 12
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
Ratio | 0.14 (0.09)

9. Secondary Outcome: Absolute Change in Drusen Area Based on Masked, Digital Grading of Fundus Photography by an External Reading Center, in the Study Eye at 12 Months Compared to Baseline.
Description: The total area occupied by drusen was determined using planimetry for color stereoscopic fundus images by masked graders at the Doheny Image Reading Center (University of Southern California, Los Angeles, CA).
  One Macular Photocoagulation Study Disc Area (MPS DA) is equivalent to 1.77 mm^2 on the retina.
Time Frame: Baseline and Month 12
Population: The analysis was intention-to-treat (ITT). Although 6 participants were enrolled, only 3 had drusen area graded at 12 months.
Measure: Mean (Standard Deviation); unit: MPS DA
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 3
Number analyzed (Eyes) | 3
MPS DA | 0.02 (0.19)

10. Secondary Outcome: Absolute Change in Drusen Area Based on Masked, Digital Grading of Fundus Photography by an External Reading Center, in the Fellow Eye at 12 Months Compared to Baseline.
Description: as for outcome 9
Time Frame: Baseline and Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: MPS DA
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 3
Number analyzed (Eyes) | 3
MPS DA | 0.29 (0.78)

11. Secondary Outcome: Absolute Change in Area of GA, as Measured by Fundus Autofluorescence (FAF) Imaging Using a Modified Fundus Camera (mFC), in the Study Eye at 12 Months Compared to Baseline.
Description: Geographic atrophy (GA) is the death of photoreceptors and surrounding cells in the retina. The death of these photoreceptors results in lesions that cause vision loss. The area of GA was determined using planimetry for FAF images obtained with a mFC by masked graders at the Doheny Image Reading Center (University of Southern California, Los Angeles, CA).
  This outcome measure was calculated by subtracting the GA value for the study eye at baseline from the GA value for the study eye at Month 12.
Time Frame: Baseline and Month 12
Population: The analysis was intention-to-treat (ITT). Although 6 participants were enrolled, only 5 were followed for 12 months.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
mm^2 | 2.75 (1.83)

12. Secondary Outcome: Absolute Change in Area of GA, as Measured by Fundus Autofluorescence (FAF) Imaging Using a Modified Fundus Camera (mFC), in the Fellow Eye at 12 Months Compared to Baseline.
Description: as for outcome 11
Time Frame: Baseline and Month 12
Population: The analysis was intention-to-treat (ITT). Although 6 participants were enrolled, only 5 were followed for 12 months.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
mm^2 | 1.44 (1.17)

13. Secondary Outcome: Absolute Change in Area of GA, as Measured by Fundus Autofluorescence (FAF) Imaging Using a Confocal Scanning Laser Ophthalmoscope (SLO), in the Study Eye at 12 Months Compared to Baseline.
Description: Geographic atrophy (GA) is the death of photoreceptors and surrounding cells in the retina. The death of these photoreceptors results in lesions that cause vision loss. The area of GA was determined using planimetry for FAF images obtained with a SLO by masked graders at the Doheny Image Reading Center (University of Southern California, Los Angeles, CA).
  This outcome measure was calculated by subtracting the GA value for the study eye at baseline from the GA value for the study eye at Month 12.
Time Frame: Baseline and Month 12
Population: The analysis was intention-to-treat (ITT). Although 6 participants were enrolled, only 5 were followed for 12 months.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
mm^2 | 2.4 (0.82)

14. Secondary Outcome: Absolute Change in Area of GA, as Measured by Fundus Autofluorescence (FAF) Imaging Using a Confocal Scanning Laser Ophthalmoscope (SLO), in the Fellow Eye at 12 Months Compared to Baseline.
Description: Geographic atrophy (GA) is the death of photoreceptors and surrounding cells in the retina. The death of these photoreceptors results in lesions that cause vision loss.The area of GA was determined using planimetry for FAF images obtained with a SLO by masked graders at the Doheny Image Reading Center (University of Southern California, Los Angeles, CA).
  This outcome measure was calculated by subtracting the GA value for the study eye at baseline from the GA value for the study eye at Month 12.
Time Frame: Baseline and Month 12
Population: The analysis was intention-to-treat (ITT). Although 6 participants were enrolled, only 5 were followed for 12 months.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
mm^2 | 1.6 (0.76)

15. Secondary Outcome: Relative Change in Area of GA, as Measured by Fundus Autofluorescence (FAF) Imaging Using a Confocal Scanning Laser Ophthalmoscope (SLO), in the Study Eye at 12 Months Compared to Baseline.
Description: Geographic atrophy (GA) is the death of photoreceptors and surrounding cells in the retina. The death of these photoreceptors results in lesions that cause vision loss. The area of GA was determined using planimetry for FAF images obtained with a SLO by masked graders at the Doheny Image Reading Center (University of Southern California, Los Angeles, CA).
  This outcome measure was calculated by dividing the absolute change in the total area of GA in the study eye at 12 months by the baseline value.
Time Frame: Baseline and Month 12
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
Ratio | 0.21 (0.14)

16. Secondary Outcome: Relative Change in Area of GA, as Measured by Fundus Autofluorescence (FAF) Imaging Using a Confocal Scanning Laser Ophthalmoscope (SLO), in the Fellow Eye at 12 Months Compared to Baseline.
Description: as for outcome 15
Time Frame: Baseline and Month 12
Population: The analysis was intention-to-treat (ITT). Although 6 participants were enrolled, only 5 were followed for 12 months.
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
Ratio | 0.15 (0.10)

17. Secondary Outcome: Relative Change in Area of GA, as Measured by Fundus Autofluorescence (FAF) Imaging Using a Modified Fundus Camera (mFC), in the Study Eye at 12 Months Compared to Baseline.
Description: Geographic atrophy (GA) is the death of photoreceptors and surrounding cells in the retina. The death of these photoreceptors results in lesions that cause vision loss. The area of GA was determined using planimetry for FAF images obtained with a mFC by masked graders at the Doheny Image Reading Center (University of Southern California, Los Angeles, CA).
  This outcome measure was calculated by dividing the absolute change in the total area of GA in the study eye at 12 months by the baseline value.
Time Frame: Baseline and Month 12
Population: The analysis was intention-to-treat (ITT). Although 6 participants were enrolled, only 5 were followed for 12 months.
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
Ratio | 0.21 (0.12)

18. Secondary Outcome: Relative Change in Area of GA, as Measured by Fundus Autofluorescence (FAF) Imaging Using a Modified Fundus Camera (mFC), in the Fellow Eye at 12 Months Compared to Baseline.
Description: as for outcome 17
Time Frame: Baseline and Month 12
Population: The analysis was intention-to-treat (ITT). Although 6 participants were enrolled, only 5 were followed for 12 months.
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Eyes
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
Ratio | 0.13 (0.10)

19. Secondary Outcome: Development of Exudative Age-Related Macular Degeneration (AMD) as Measured by Optical Coherence Tomography (OCT) at 12 Months Compared to Baseline
Time Frame: Baseline and 12 Months
Population: Zero participants were analyzed because no data were collected to analyze this outcome as no study or fellow eye developed neovascular changes during the study.
Arm/Group | Sirolimus
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Sirolimus
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=6)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Heart valve incompetence (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=6)
Age-related macular degeneration (Eye disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Basophil count decreased (Investigations) | 1 (1)
Blood alkaline phosphatase decreased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Blood calcium decreased (Investigations) | 1 (1)
Blood glucose abnormal (Investigations) | 3 (3)
Blood urea increased (Investigations) | 2 (2)
Bone density abnormal (Investigations) | 1 (1)
Full blood count abnormal (Investigations) | 1 (1)
Haematocrit decreased (Investigations) | 1 (1)
Haemoglobin urine present (Investigations) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Lipids decreased (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Monocyte count abnormal (Investigations) | 1 (1)
Monocyte count decreased (Investigations) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Ocular discomfort (Eye disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 1 (1)
Red blood cell count increased (Investigations) | 1 (1)
Red blood cells urine (Investigations) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin lesion excision (Surgical and medical procedures) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Visual acuity reduced (Eye disorders) | 1 (1)
Lipids increased (Investigations) | 1 (1)
Mild pain (General disorders) | 1 (1) — Verbatim adverse event description

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No